CLINICAL TRIAL: NCT04615000
Title: SeroCovid<19: A Prospective Covid-19 Seroconversion Study in a Tertiary Pediatric Patient Cohort
Brief Title: SeroCovid<19: Covid-19 Seroconversion in Tertiary Pediatric Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-08104
Record Dates: First submitted 2020-11-03; First posted 2020-11-04 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Children, Only
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 serological assessment (IgG) — Periodic assessment of the serology status (SARS-CoV-2 specific IgG) with a 3 to 6 month interval

SUMMARY:
Children are relatively spared from the direct clinical impact of COVID-19. Pediatric patients with regular follow-up at tertiary pediatric centres and presenting one or more chronic conditions might be at increased risk for severe COVID-19. With a prospective seroprevalence study, we aim to study COVID-19 incidence, disease course and risk factors associated with SARS-CoV-2 infection in this specific context.

DETAILED DESCRIPTION:
Children and adolescents seem to be relatively spared from severe SARS-CoV-2 infection. Throughout the course of the COVID-19 pandemic, these findings were confirmed with, for example, also in Belgium only 1.8% of the confirmed infections, 1.6% of the hospitalizations in intensive care, and 0.011% of the deaths from COVID-19 attributed to children by the end of May 2020. Multiple immunological hypotheses (ACE2 expression, lymphocyte repertoire, cross immunization) have been suggested without one clear explanation to date. In addition, children seem to play a limited role in the spread of the virus and are not considered the "engine of the epidemic".

Population seroconversion studies have been initiated with the determination of antibodies to SARS-CoV-2. For Belgium, seroconversion rates were estimated at around 2.1% at the end of March, 4.3% in mid-April, 6% at the beginning of May and 6.9% at the end of May 2020, comparable to international studies. However, even with these prospective studies, it remained unclear whether the seroconversion rate in children is comparable to adults. In addition, it has not yet been demonstrated whether the mild course and limited hospitalizations in children are related to either a mild course or (in part) also to a lack of exposure to SARS-CoV-2 and therefore limited seroconversion in children.

With this study we aim to monitor both the presence of antibodies (serology) in children with chronic disease, followed in a tertiary hospital in Belgium, combined with the registration of the clinical course of COVID-19 in this population. In addition, we want to correlate the social activities with the risk of exposure to the virus and subsequent seroconversion. Blood samples for serology are performed at a 3- to 6-month interval, linked to an already planned blood sample for diagnostic reasons. This data will allow to gain more insight into the actual rate of infection and the symptoms caused by COVID-19 in children with a chronic disease, on the one hand, and, on the other hand, how the social behavior, limited by the lockdown measures or after its progressive relaxation, affects seroconversion in these pediatric populations. These data may or may not confirm current hypotheses about infection rate and clinic severity and will also influence current and future policies such as closing schools and defining at-risk populations.

ELIGIBILITY:
Inclusion Criteria:

* children <18 years of age
* a clearly defined chronic condition requiring follow-up at the tertiary pediatric hospital of the Ghent University Hospital
* routine blood sampling planned per 3 to 6 months

Exclusion Criteria:

* no clear diagnosis or reason for follow-up at the Ghent University Hospital
* no routine blood sampling planned
* unable to understand or provide informed consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * children <18 years of age
  * a clearly defined chronic condition requiring follow-up at the tertiary pediatric hospital of the Ghent University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate of children with chronic conditions followed in a tertiary centre | 12-18 months
  Prospective follow-up of the COVID-19 seroconversion rate (serum IgG) of children with chronic conditions followed in a tertiary centre

SECONDARY OUTCOMES:
Epidemiological and social determinants of SARS-CoV-2 infection risk in children with chronic conditions | 12-18 months
  Questionnaire assessment of the epidemiological (household, school,... infections) and social determinants (school, daycare, sport participation,...) of SARS-CoV-2 infection risk in children with chronic conditions
Clinical manifestations of COVID-19 in children with chronic conditions | 12-18 months
  Questionnaire assessment of COVID-19 associated symptoms in the subcohort of patients with seroconversion

CONTACTS AND LOCATIONS:
Overall Officials: Filomeen Haerynck, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided